CLINICAL TRIAL: NCT05326009
Title: A Direct Comparative Study of Tau Tracer in Patients With Alzheimer's Disease
Acronym: HTH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: H. Lundbeck A/S (Industry); Hoffmann-La Roche (Industry); Genentech, Inc. (Industry); Life Molecular Imaging SA (Industry); APRINOIA Therapeutics (Industry); XINGIMAGING LLC (Unknown); Hangzhou G-Bio Biotechnology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Piu Chan, Professor, Xuanwu Hospital, Beijing
Other Study IDs: 104
Record Dates: First submitted 2022-02-17; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheier Disease; PET imaging; AV45; AV1451; Tau
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — venous blood collected with EDTA anticoagulant CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, a total of 60 AD patients with Aβ deposition will beenrolled.Qualified subjects will complete PET imaging scan of Tau imaging agent inXuanwuHospital, and each subject will receive three of the following five imaging agents: PI-2620, APN1607, AV1451, RO948 or GTP1.The imaging time interval between the two tracers should be at least 4 days but less than 4 weeks. All PET scans of each subject were completed within 3 months.To compare the different Tau tracers' binding ability (SUVR or Tau distribution change) of the same subject in AD population. Obtain the safety data of each tracer after injection.

DETAILED DESCRIPTION:
Patients with AD in prodromal stage, mild or moderate degree, who have stable medical condition and meet the inclusion criteria, do not meet any exclusion criteria, will be eligible for inclusion in this study.

[18F] florbetapir PET imaging will be used to evaluate amyloid deposition during the screening period. If [18F] florbetapir imaging confirmed amyloid deposition based on positive visual reading and SUVR > 1.1, the patient was considered to be amyloid deposition positive.After the subjects enter the group, the comprehensive collection of clinical information, the assessment of cognitive related scale and the collection and detection of biological samples are carried out. Qualified subjects will complete PET imaging scan of Tau imaging agent in Xuanwu Hospital, and each subject will receive three of the following five imaging agents: PI-2620, APN1607, AV1451, RO948 or GTP1. All subjects will sign the tracer related informed consent before PET tracer injection. Imaging will be carried out as detailed in the technical operation manual. PET center staff will closely observe and evaluate adverse events of subjects throughout the process, and allow them to leave the hospital after confirming medical stability. After 48 hours of scanning, the staff will follow up the subjects by telephone to confirm the health status of the subjects and record the information related to adverse events. The imaging time interval between the two tracers should be at least 4 days but less than 4 weeks. All PET scans of each subject were completed within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-80, male or female.
* The legal authorizer or caregiver of the subject (if applicable) needs to sign the informed consent before any assessment.
* Based on the NINCDS / ADRDA and DSM-IV standards, it is likely to have AD dementia, with mild severe amnesia.
* Screening CDR score = 0.5, and MMSE score is between 24-26 (AD patients in prodromal stage).
* Or,
* CDR score = 0.5 or 1, and MMSE score is between 20-23 (mild AD patients) -Or,
* CDR score = 2, and MMSE score is between 15-21 (for moderate AD patients).
* It has received PET imaging examination of amyloid protein or [18F] florbetapir imaging examination within 12 months before screening, and it is confirmed that there is amyloid binding based on qualitative analysis (visual read) and quantitative analysis. The results of amyloid PET imaging will be shared with participants, and the scanning results may be used by participants for future research.
* There is no obvious evidence of other neuropathology in brain MRI supporting AD diagnosis.
* Before the screening visit date, patients taking symptomatic treatment drugs must maintain a stable maintenance dose for at least 30 days.
* Female subjects must have medical records or doctor's records for surgical infertility (through hysterectomy, bilateral ovariectomy or tubal ligation) or at least 1 year after menopause, otherwise, pregnancy test is required in screening period and every scanning visit and should be negative. Male subjects and their fertile partners must promise to use two methods of contraception during the study period, and one of them is barrier contraception for male subjects.
* Male subjects are not allowed to donate sperm during the study and within 90 days after the completion of the study.
* Willing and able to cooperate with the research process.
* A qualified subject's Research Companion needs regular and sufficient contact between the research companion and the subject (weekly time ≥ 10 hours), can provide accurate information about the subject's cognition and function, and agrees to accompany the subject and provide relevant information during the visit. The study companion must have sufficient cognitive ability to accurately report the behavior, cognition and function of the subjects. The same study companion should be able to accompany the subjects to participate in the whole study process.

Exclusion Criteria:

* Any existing or 3-year history of alcohol or drug abuse (self statement)
* Laboratory examination or ECG indicates significant clinical abnormalities and / or important unstable clinical diseases.
* In the past year, the amount of radiation received by participating or clinical clinics in combination with this research institute has exceeded 50mSV (the annual limit allowed by FDA for research volunteers).
* Serious gastrointestinal, cardiovascular, liver and kidney, blood, tumor, endocrine, potential nervous system, immune deficiency (including HIV positive), pneumonia and other diseases. Stable, treated chronic disease conditions such as high blood pressure, hyperlipidemia, diabetes, non metastatic skin cancer or prostate cancer, which researchers believe will not cause cognitive impairment or restrict participation in the study, are acceptable.
* In addition to AD, the history or current status of neurological diseases that may affect cognition, including but not limited to Parkinson's disease, cortical basal ganglia degeneration, dementia of Lewy body, CJD, Huntington's disease, normal intracranial pressure hydrocephalus, tic disease, hypoxia, or other serious CNS trauma with significant clinical significance.
* Other diseases or causes may cause the subjects to fail to complete the whole study.
* MRI exclusion criteria include: evidence that may affect cognition, such as significant evidence of cerebrovascular disease (more than two lacunar infarcts, any infarct larger than 1cm3, or deep white matter abnormality, equivalent to Fazekas score level 3, at least one fusion high signal lesion on FLAIR sequence, i.e. ≥20mm in any dimension), infectious diseases, space occupying lesions, normal pressure hydrocephalus, central nervous system injury or any other structural abnormality that may affect cognition.
* Internal implants such as cardiac pacemaker or defibrillator, insulin pump, cochlear implant, metal eye foreign body, implanted nerve stimulator, central nervous system aneurysm clip and other medical implants that can not receive MRI, or MRI examination has a history of claustrophobia.
* Daily use of anticholinergic antidepressants, typical antipsychotics or barbiturates. Infrequent use of typical antipsychotics for vomiting or barbiturates for migraine treatment is permitted, provided that no dose is taken during the 5 half lives prior to screening or any neurocognitive assessment.
* Daily use of benzodiazepines, opioids or opioids. However, intermittent short-term treatment is permitted, except for use in the 5 half-lives prior to screening or any neurocognitive assessment.
* Use hypnotics, stimulants, atypical antipsychotics, central anticholinergic antihistamines, or anticholinergic antispasmodics with central effect, unless (a) they are administered daily, so that they will not start or stop treatment or dose change within the first five half lives of screening or at any time during the study period, or (b) they are administered intermittently and in a short period, while in screening or neurocognition Not used in the first 5 half lives of the assessment.
* In the 12 months before screening, use any therapeutic molecule or treatment method targeting Aβ, or use the treatment targeting tau in the 24 months before screening

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, a total of 60 AD patients with Aβ deposition will be enrolled.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
To compare the different Tau tracers' binding ability of the same subject in AD population. | August 2021 to May 2023
  SUVR value was used to compare AD population different Tau targeting tracers, evaluate the tau binding capacity of different Tau tracers in AD population,
Assessing the potential value of tracers in AD diagnosis | August 2021 to May 2023
  Comparison of specific regions bound to specific tau tracers in the same subject AD population at each visit
To compare the different Tau tracers' binding ability of the same subject in AD | August 2021 to May 2023
  Tau distribution changewas used to compare AD population different Tau targeting tracers, evaluate the tau binding capacity of different Tau tracers in AD population
Obtain the safety data of each tracer after injection. | August 2021 to May 2023
  Number of adverse events recorded from baseline to follow-up by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Biao Chen, Doctor, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No